CLINICAL TRIAL: NCT07214077
Title: Harmonized Healing: Personalized Music Interventions to Address Chronic Pain in People Living With HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Fenway Institute (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Peter R Chai MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P002274
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Hiv
Keywords: Chronic Pain; Music; smartphone app
MeSH Terms: conditions — Chronic Pain; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harmonized Healing App (Experimental): Participants will receive psychoeducation related to drivers of chronic pain in the context of HIV and tips for managing pain, and the Harmonized Healing app. Participants will use the app at least once daily, or as needed, to manage and alleviate pain exacerbations for 3 months.
  Interventions: Behavioral: Harmonized Healing App; Behavioral: Psychoeducation
- Control (Active Comparator): Participants will receive psychoeducation related to drivers of chronic pain in the context of HIV and tips for managing pain. Participants will review the information at least once before each monthly visit (Month 1 to 3 Visits).
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Harmonized Healing App — A smartphone-driven music-based intervention designed to support daily or as-needed use of personalized music to manage and alleviate pain exacerbations.
  Arms: Harmonized Healing App
Behavioral: Psychoeducation — Educational materials on drivers of chronic pain in the context of HIV and strategies for pain management.

SUMMARY:
The goal of this randomized controlled trial is to understand the feasibility and acceptability of a music-based mobile application to address chronic pain in people with HIV. Participants in the intervention group will use the Harmonized Healing music app daily, or as needed, for 3 months. Participants in the control group will receive psychoeducation on chronic pain and strategies for pain management. All participants will attend monthly follow-up visits during the 3-month intervention period, and an additional follow-up visit at Month 6.

DETAILED DESCRIPTION:
Harmonized Healing is a novel, smartphone-driven, music-based behavioral intervention designed to help manage chronic pain in people with HIV. This two-arm pilot randomized controlled trial will enroll 60 individuals living with HIV and chronic pain. Participants will be randomized to receive either Harmonized Healing plus psychoeducation (intervention arm) or psychoeducation alone (control arm). Those in the intervention arm will be asked to use the Harmonized Healing music app daily, or as needed, for 3 months. Participants in both groups will attend monthly study visits during the 3-month intervention period, and one additional follow-up visit at Month 6.

The primary objective of this pilot study is to evaluate the feasibility and acceptability of the Harmonized Healing app. In addition, qualitative feedback will be collected from participants who used Harmonized Healing to better understand their experiences with the intervention and participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Owns a smartphone
* Living with HIV
* Currently prescribed antiretroviral therapy (ART) for HIV
* Experience with chronic pain (determined by self-reported pain of ≥3 on the Brief Pain Inventory for at least 3 months)

Exclusion Criteria:

* Have a significant hearing loss
* HIV-negative
* Have been prescribed naltrexone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility: Recruitment | Month 3 Study Visits
  Intervention feasibility will be assessed by the proportion of eligible individuals from the available recruitment pool.
Intervention Feasibility: Enrollment | Month 3 Study Visits
  Intervention feasibility will be assessed by the proportion of eligible individuals who consent and enroll, and the proportion of the target sample size achieved.
Intervention Feasibility: Attrition | Month 3 and Month 6 Study Visits
  Intervention feasibility will be assessed by the proportion of participants retained at each follow-up visit.
Intervention Feasibility: Adherence to Assessment Battery | Month 3 and Month 6 Study Visits
  Intervention feasibility will be assessed by the proportion of participants who completed the assessment battery at each study visit. In the intervention condition, this includes the proportion of EMA completion.
Intervention Feasibility: FIM | Month 3 Study Visit
  The Feasibility of Intervention Measure (FIM) is a 4-item Likert feasibility scale ranging from 1 (Completely disagree) to 5 (Completely agree). A mean score is calculated, resulting in a continuous score with higher scores indicating greater intervention feasibility.
Intervention Acceptability: Fidelity | Month 3 Study Visit
  Intervention fidelity will be assessed by adherence to assigned study activities. In the intervention arm, this includes the proportion of days adherent to the prescribed app use. In the control arm, this includes the proportion of psychoeducation reviews completed before monthly visits.
Intervention Acceptability: Engagement (Percentage of days used) | Month 3 Study Visit
  Intervention engagement will be assessed by the proportion of days with app use.
Intervention Acceptability: Engagement (Minutes engaged per week) | Month 3 Study Visit
  Intervention engagement will be assessed by minutes of app engagement per week.
Intervention Acceptability: AIM | Month 3 Study Visit
  The Acceptability of Intervention Measure (AIM) is a 4-item Likert agreeability scale ranging from 1 (Completely disagree) to 5 (Completely agree). A mean score is calculated, resulting in a continuous score with higher scores indicating greater intervention acceptability.
Intervention Acceptability: Qualitative Exit Interviews | Month 3 Study Visit
  Intervention acceptability will be assessed via qualitative interviews exploring participants' lived experiences using the Harmonized Healing app, including facilitators and barriers to use, and engagement with the app.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chai, MD, MMS, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Identifying information may be redacted and data shared based on reasonable request from researchers.